CLINICAL TRIAL: NCT03191539
Title: Assessment of the Clinical and Ultrasound Response to Apremilast by Clinical Evaluation and by a Joint-periarticular-nail Ultrasound Index in Patients With Active Psoriatic Arthritis
Acronym: APREMILAST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSA-PI-006421
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-06

CONDITIONS: Arthritis; Psoriasis (Etiology)
MeSH Terms: conditions — Arthritis; Psoriasis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apremilast (Experimental): 30 mg of Apremilast twice a day during 52 weeks. During the first 6 days will be a dose escalation as the following: Day 1: 10 mg daily Day 2: 10 mg day- 10 mg night Day 3: 10 mg day- 20 mg night Day 4: 20mg day- 20mg night Day 5: 20 mg day- 30 mg night Day 6: 30 mg day- 30 mg night
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — 30 mg twice a day during 52 weeks. In the first 6 days will be a dose escalation

SUMMARY:
This study aims to evaluate more objectively, through an imaging technique such as ultrasound, changes in joints and entheses of patients with active psoriatic arthritis (PAs) who will start treatment with Apremilast after the failure of other therapies such as synthetic DMARD (metrotrexato , Leflunomide ...).

The hypothesis of the study is that the technique of ultrasound can demonstrate the efficacy of Apremilast in the treatment of patients with active PAs

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older with Psoriatic Arthritis (PsA) according to Classification Criteria for Psoriatic Arthritis (CASPAR) criteria at the time of selection, with involvement of hands and/or feet with active clinical disease (more than two swollen joints)
* Present 2 or more joints with ultrasound synovitis at the screening visit
* Present 1 or more entheses affected as shown by ultrasound at the screening visit
* Accept and sign the informed consent of the study
* Ability to comply with all tests and visits of specified protocol and have a permanent address.
* Women of childbearing potential must have a negative pregnancy test at the baseline visit. Women of childbearing potential who participate in the study should use one of the following contraceptive methods throughout the trial and for at least 28 days after taking the last dose of study medication.
* Approved contraceptive options are:

Option 1: Any of the following: hormonal contraceptives (e.g., birth control pills, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or her partner has had a vasectomy OR Option 2: Male or female condom (a latex condom or non-latex condom but NOT made of natural membrane [animal, e.g., polyurethane]) AND one of the following additional barrier methods: a) diaphragm with spermicide; B) cervical cap with spermicide; or c) contraceptive sponge with spermicide.

Exclusion Criteria:

* Concomitant treatment with methotrexate or leflunomide or other DMARDs. Patients may not have taken methotrexate during the month prior to screening, leflunomide during the 2 months prior to screening and other DMARDs during the 15 days prior to screening
* Prior or current use of biological therapy (anti-TNF)
* Failure to meet any of the inclusion requirements
* Medical contraindications for taking Apremilast
* Pregnancy or breastfeeding
* History of allergy to any component of the study drug
* Active tuberculosis (TB) or history of incomplete treatment for tuberculosis
* Substance abuse or history of substance abuse within 6 months prior to screening
* Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks prior to screening
* Malignancy or history of malignancy (except in situ basal or squamous cell skin carcinomas treated [i.e., cured] and treated cervical intraepithelial neoplasms [i.e., cured] or carcinoma in situ of the cervix without evidence of recurrence within the last 5 years)
* Use of systemic corticosteroids at doses >10 mg/day at the time of screening and 4 weeks before
* Use of potent cytochrome CYP3A4 enzyme inducers (e.g., rifampicin, phenobarbital, carbamazepine, phenytoin, St. John's wort and grapefruit juice) at the time of screening, 4 weeks before or during the study
* Use of phototherapy within 4 weeks prior to screening (i.e., Ultraviolet B (UVB), psoralen and ultraviolet A (PUVA))
* Use of any investigational drug within 4 weeks prior to screening
* Prior treatment with Apremilast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-11-02 (Estimated); Primary Completion 2019-06-14 (Estimated); Study Completion 2019-06-14 (Estimated)

PRIMARY OUTCOMES:
Reduction in the ultrasound index | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months
  Reduction in the ultrasound index at 12 months after the introduction of Apremilast in the study patients

SECONDARY OUTCOMES:
Disease Activity Score (DAS 28) | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months
Psoriasis activity and severity index (PASI) | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months
Leeds Enthesitis Index (LEI) | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months
Number of tender and swollen joints assessed by (Number of Tender Joints (NTJ) ) | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months
Patient Visual Analog Scale (VAS) for pain | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months
Ultrasonic nail injuries | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months
Clinical Disease Activity Index (CDAI) | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months
Simple Disease Activity Index (SDAI) | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months
Number of tender and swollen joints assessed by (Number os swollen joints (NSJ)) | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months
doctor Visual Analog Scale (VAS) for pain | screening visit, baseline visit, visit 1 month, visit 6 months, visit 9 months and visit 12 months

IPD SHARING:
Plan to Share IPD: No